CLINICAL TRIAL: NCT01192555
Title: A Phase I/II Study Using Allogeneic Tumor Cell Vaccination With Oral Metronomic Cytoxan in Patients With High-Risk Neuroblastoma (ATOMIC)
Brief Title: Allogeneic Tumor Cell Vaccination With Oral Metronomic Cytoxan in Patients With High-Risk Neuroblastoma
Acronym: ATOMIC
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Malcolm Brenner, Principal Investigator, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-26652-ATOMIC
Record Dates: First submitted 2010-08-16; First posted 2010-09-01 (Estimated); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; Chemotherapy; Pediatrics; Cytoxan; immunotherapy; vaccine
MeSH Terms: conditions — Neuroblastoma | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Plan (Experimental): Neuroblastoma Vaccine (unmodified SKNLP, with gene-modified SJNB-JF-IL2 and SJNB-JF-LTN neuroblastoma cells) and Cytoxan (Cyclophosphamide)
  Interventions: Biological: Neuroblastoma Vaccine (unmodified SKNLP, with gene-modified SJNB-JF-IL2 and SJNB-JF-LTN neuroblastoma cells; Drug: Cytoxan

INTERVENTIONS:
Biological: Neuroblastoma Vaccine (unmodified SKNLP, with gene-modified SJNB-JF-IL2 and SJNB-JF-LTN neuroblastoma cells — 1x10^7cells/m2 each of unmodified SKNLP, with gene-modified SJNB-JF-IL2 and SJNB-JF-LTN neuroblastoma cells will be given by subcutaneous injection while suspended in Ringers solution with 5% HSA in a single syringe in a volume of up to 1 ml.
  Vaccines will be given on day 0 of week 0 and then on day 0 (+ 72 hours) of weeks 2, 4, 6, 9, 12, 16, 20.
  Cells will be administered as a subcutaneous injection over 1 minute using a 21-gauge needle. Procedural pain control methods may be used per institutional protocol.
  Other Names: SKNLP w/ gene-mod. SJNB-JF-IL2 & SJNB-JF-LTN neurobl. cells
Drug: Cytoxan — Metronomic oral cytoxan will start 72 hours prior to the first vaccination at a dose of 50 mg/m2/day. Cytoxan will be held on the day of vaccine administration and for the next 96 hours. After the first vaccine, patients will take 25 mg/m2/day as outlined on the roadmap.
  Other Names: Cyclophosphamide

SUMMARY:
Neuroblastoma is the second most common solid tumor seen in children, but causes approximately 15% of childhood cancer deaths each year. Patients with high-risk disease require treatment with a combination of chemotherapy, surgery, radiation, and stem cell transplant; however, many will have their disease come back within 3 years. Due to this high rate of relapse, this study is being done to investigate an experimental treatment option for children whose disease has returned.

This clinical trial is for patients with neuroblastoma that has either come back after treatment or never went away in the first place. A series of immunizations will be administered using a tumor vaccine and add low-dose chemotherapy to be taken by mouth on a daily basis. The hope is that the vaccine will cause the immune system to recognize and kill more types of neuroblastoma tumors. Additionally, the immunizations will be combined with daily low dose chemotherapy. Daily low-dose chemotherapy, also know as metronomic chemotherapy, works by attacking the blood vessels that allow tumors to grow. Using metronomic doses of a drug called cytoxan can also decrease T regulatory cells, a specific type of cell that tumors use to hide from the immune system.

The purpose of this study is to test the safety and anti-tumor effect of the tumor cell vaccination plus low dose, metronomic chemotherapy in treating patients with relapsed/refractory neuroblastoma.

DETAILED DESCRIPTION:
WHAT IS THE OVERALL TREATMENT PLAN AND HOW MANY VACCINATIONS WILL THE PATIENT RECEIVE? There will be several injections of the vaccine scheduled. The first injection will be given 3 days after starting oral cytoxan. The 2nd to 4th injections will be given approximately every 14 days after the previous vaccine. During this time, the patient will be taking oral cytoxan once a day except on the day of and 4 days following the vaccine. Two to 3 weeks after the 4th vaccine, the patient will have a complete evaluation of their disease. If the scans and lab tests show that the patient has not had any serious side-effects, they will be eligible to receive 4 additional vaccinations given at 3 week intervals. The disease will be re-evaluated again after vaccine numbers 6 and 8. If the patient is able to complete the entire study, they will have received a total of 8 vaccinations and the last dose of oral cytoxan will be 1 month after the 8th vaccination. Total time duration for participating in this study is 15 years (treatment portion within year 1 and follow up during years 2-15).

Neuroblastoma vaccinations are given like many other vaccines. They will be given subcutaneously. The injections will be 1/10th of a teaspoon.

MEDICAL TESTS BEFORE STARTING TREATMENT:

Before starting low dose chemotherapy plus oral cytoxan, patients will receive a series of standard medical tests:

* Physical exam
* Blood tests to measure blood cells, blood salts, kidney and liver function
* Measurements of their disease (CT or MRI of the primary tumor site and any locations of tumor spread; MIBG or Bone scan; Chest X-ray if they did not have a CT of the chest; and bone marrow studies if the patient has known bone marrow disease)
* Baseline testing of immune function
* Pregnancy testing will be performed on females of child bearing age

MEDICAL TESTS DURING AND AFTER TREATMENT:

Prior to each vaccine dose, the patient will receive:

* Physical exam
* Blood tests to measure blood cells, blood salts, kidney and liver function
* Measurements of the disease (CT or MRI of the primary tumor site and any locations of tumor spread; MIBG or Bone scan; Chest X-ray if they did not have a CT of the chest; and bone marrow studies if they have known bone marrow disease) after the 4th, 6th and 8th vaccine.
* Testing of immune function
* Pregnancy testing will be performed again on females of child bearing age prior to the 5th vaccine

To learn more about the way the vaccine is stimulating the immune cells, we will collect blood prior to each vaccination and at scheduled time points until 3 months after the last vaccine treatment. The total amount of blood to be collected on any day is no more than 2 ounces, but will depend upon the weight. This volume is considered safe in teens and adults, but may be decreased if the patient is anemic. On days when the patient receives the vaccine, blood will be taken before the cells are given.

ELIGIBILITY:
INCLUSION CRITERIA:

* Histologically proven high risk neuroblastoma in first or subsequent relapse or with primary refractory disease or inability to complete standard therapy
* Age less than 21 at time of initial diagnosis
* Life expectancy 12 weeks or greater
* Karnofsky or Lansky score of 50 or greater
* Platelet count of 50,000/ul or greater
* ANC greater than 750/ul
* Alk Phos level less than 2.5 x upper limit of normal
* Bilirubin less than 2x normal
* AST less than 3x normal
* Hgb 8.0 or greater
* Creatinine 2 x ULN or less OR GFR greater than 40 ml/min/1.73 m2
* Patient has recovered from last chemotherapy or investigational therapy prior to study enrollment
* Women of child-bearing potential must not be pregnant and take/use effective birth control while participating in the study.

EXCLUSION CRITERIA:

* Due to the unknown effects of this therapy on a fetus, pregnant women will be excluded from this research
* Women who are breast-feeding
* Known HIV positive subjects since treatment may be immunosuppressive
* Severe intercurrent infection or uncontrolled condition including, but not limited to ongoing or active infection, symptomatic heart failure, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Previous use of oral cytoxan for more than 2 consecutive months within the last 6 months
* Patients currently receiving any investigational agents or have received any tumor vaccines within the previous six months
* Patients, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-09; Primary Completion 2012-07 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | week 30
  Phase I Primary Objective: Evaluate the safety of fixed dose oral cytoxan administered metronomically to coincide with repeated immunizations of gene-modified, IL-2/lymphotactin secreting SJNB-JF-IL2 and SJNB-JF-LTN cells co-administered with unmodified SKNLP neuroblastoma cell lines in patients with a history of relapsed/refractory high-risk neuroblastoma.

SECONDARY OUTCOMES:
Participants with T-cell changes as a Measure of Immune Response | 15 years
  Phase I Secondary Objective: Evaluate the immune response to combination metronomic chemotherapy and allogeneic tumor cell immunizations.
Number of Participants with Disease Progression as a Measure of Efficacy | 10 weeks
  Phase II Primary Objective: Evaluate time to progression after administration of combination metronomic chemotherapy and allogeneic tumor cell immunizations in patients with a history of relapsed/refractory high-risk neuroblastoma.

OTHER OUTCOMES:
Analysis of Immunologic Measurements | 15 years
  Phase II Secondary Objectives:
  1. Evaluate changes in T regulatory cell absolute number, percentages, and suppressive function after the use of metronomic low-dose oral cytoxan with allogeneic neuroblastoma tumor cell immunizations.
  2. Evaluate the alterations in angiogenic biomarkers related to fixed dose oral cytoxan and repeated immunizations with allogeneic tumor cell immunizations.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Brenner, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States